CLINICAL TRIAL: NCT05842603
Title: I Can Move With Purpose Now! A Pilot Lifestyle Intervention Study in Myeloproliferative Neoplasm Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gabriela Hobbs, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-692
Record Dates: First submitted 2023-04-10; First posted 2023-05-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Myeloproliferative Disorders; Leukemia
Keywords: Myeloproliferative Disorders; Leukemia
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiac Lifestyle Program (Experimental): Participants will complete study procedures as follows:
  * Baseline in-clinic visit with research team doctor for history and physical and the completion of questionnaires.
  * 6 virtual group classes alternating with 6 in-person group classes.
  * Semi-structured exit interview.
  Interventions: Behavioral: Cardiac Lifestyle Program

INTERVENTIONS:
Behavioral: Cardiac Lifestyle Program — 12-week, tailored nutrition and physical activity program comprised of virtual and in-person classes.

SUMMARY:
The goal of this study is to see if patients with myeloproliferative disorders are able to successfully complete the Cardiac Lifestyle Program(CLP). The goal of the CLP is to teach patients how to become more active and eat healthier foods.

The name of the intervention used in this research study is:

Cardiac Lifestyle Program (a 12-week, tailored nutrition and physical activity program)

DETAILED DESCRIPTION:
This is a single-arm, prospective pilot study that will enroll eligible Myeloproliferative Neoplasms (MPN) patients in a 12-week exercise and nutrition-based Cardiac Lifestyle Program (CLP). This research study is a Feasibility Study, which is the first time investigators are examining this exercise program in myeloproliferative disorder patients.

Study procedures include screening for eligibility, an in-clinic visit, questionnaires, program group classes, and blood work.

Participation in this research study is expected to last 12 weeks.

It is expected that about 30 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

-≥18 years of age

* Diagnosed with an MPN by WHO 2016 criteria,22 including essential thrombocythemia (ET), polycythemia vera (PV), prefibrotic myelofibrosis (pre-MF), myelofibrosis (MF), and MPN not otherwise specified (NOS). Within MF patients, only patients who are low or intermediate-1 risk by the Dynamic International Prognostic Scoring System (DIPSS) are eligible.23 All risk groups are eligible for the remaining MPN subtypes.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Must have at least one cardiovascular risk factor including: Body mass index (BMI) >25 kg/m2, hypertension, hyperlipidemia, diabetes mellitus or pre-diabetes or metabolic syndrome, or any prior history of cardiovascular disease, transient ischemic attack, stroke, or peripheral vascular disease. Patients not meeting any cardiovascular risk criteria must receive prior approval from the PI to participate in this study.

Exclusion Criteria:

-- MF patients with intermediate-2 or high-risk disease by DIPSS

* ECOG performance status >2.
* Any injury or medical condition that would prohibit being able to safely perform exercise, as determined by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants that Complete at Least 9 Weeks of the 12 week Program | Enrollment to end of the 3 month follow-up of last patient enrolled
  Feasibility of this pilot trial will be measured by the number of participants that complete at least 9 weeks of the exercise program. This trial will be considered feasible if at least 70% (≥21) of participants complete the program. Completion rates will be measured with a 95% confidence interval for the adherence proportion calculated by exact binomial method.

SECONDARY OUTCOMES:
Change in MPN SAF-TSS Score from Baseline to Week 12 | Baseline and Week 12 (end of program completion)
  The MPN-SAF TSS is a validated 10-item symptom assessment form that captures the most common symptoms affecting MPN patients, and is considered a standard assessment in clinical trials evaluating interventions in MPN patients. Possible scores range from 0 to 100. Change = Week 12 Score - Baseline Score.
Change in FACIT-Fatigue Score from Baseline to Week 12 | Baseline and Week 12 (end of program completion)
  The FACIT-F is a 41-item questionnaire consisting of the FACT-G (28 items), which measures health-related quality of life covering four domains of well-being (physical, social/family, emotional, functional), plus 13 fatigue-specific items. Possible scores range from 0 to 164. Change = Week 12 Score - Baseline Score.
Change in HADS Score from Baseline to Week 12 | Baseline and Week 12 (end of program completion)
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-report measure of depressive and anxiety symptoms specifically designed for use with medical patients. Possible scores range from 0-42. Change = Week 12 Score - Baseline Score.
Change in IPAQ Short Form Score from Baseline to Week 12 | Baseline and Week 12 (end of program completion)
  The IPAQ Short Form is a 7-item questionnaire that measures the amount and time spent doing various levels of physical activity over the last week. Participant answers are based on number of minutes, hours, or days spent on performing activities of various intensities. Change = Week 12 scores on each item - Baseline scores on each item.
Changes in Healthy Eating Index (HEI) Score from Baseline to Week 12 | Baseline and Week 12 (end of program completion)
  The Automated Self-Administered Dietary Assessment Tool (ASA24), a free web-based 24-hour dietary recall tool developed by the National Cancer Institute. Responses will be used to calculate a Healthy Eating Index (HEI) score, which is based on density values/ratios of intake per total energy. The HEI is a measure of dietary quality that addresses compliance with the 2015 USDA dietary guidelines. Change = Week 12 scores - Baseline scores.
Hematologic Response Rate | Baseline and Week 12 (end of program completion)
  Hematologic response rates are defined by International Working Group (IWG) working criteria including proportion of patients achieving all of the following: platelet count ≤ 400 x 109/L, WBC count <10 x 109/L, and absence of leukoerythroblastosis, hematocrit <45%.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Hobbs, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation.